CLINICAL TRIAL: NCT04591353
Title: A Randomized-controlled, Double-blind, Single-center Trial Comparing Impact of PENG Block on Quality of Recovery Compared to No-block for Primary Total Hip Arthroplasty
Brief Title: Trial Comparing Impact of PENG Block on Quality of Recovery Compared to No-block for Primary Total Hip Arthroplasty
Acronym: (PENG)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Promil Kukreja, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-300006163
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-07

CONDITIONS: Total Hip Arthroplasty
Keywords: PENG; THA; nerve blocks
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Upon enrollment in the study, participants will be randomized 1:1 to either the investigational group ("PENG Block" group) or the control group ("No Block" group). Participants will be randomized using a random number generator. The randomization will be performed using computer-generated random numbers. The study will follow a 1:1 allocation ratio for the intervention (PENG) and control (No-PENG). A random permuted block will be used to reduce the predictability of allocation. The randomization sequence will be generated using computer software using a block randomization method where blocks are variable in size (minimum block size four). The study will use a sealed opaque envelope as method to comply with allocation concealment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Investigational group ("PENG Block" group) (Experimental): Participants in the pericapsular nerve group block (PENG) arm will receive a PENG block preoperatively in the block area placed under direct ultrasound guidance as follows: Parenteral midazolam and fentanyl will be titrated to patient comfort. Standard skin sterilization, prepping and draping will be applied to the area Anatomical landmarks identified using ultrasound and skin will be numbed using 2-3 cc of 2% lidocaine. Long acting local anesthetic, a bolus of 25 cc of 0.5 % Bupivacaine will be injected lateral to iliopubic eminence (IPE). A Curvilinear low frequency (2-5 MHz) ultrasound probe will be used to identify landmarks. A 22 G, 10 cm needle will be inserted using in-plane technique and advanced to target site (17).
  Interventions: Drug: PENG Block
- Control group (Active Comparator): Control group participants will be transferred to the block area preoperatively, and care will proceed as if they were receiving injection.
  Patients will be placed in the supine position resting comfortably. Standard noninvasive monitors will be applied, and oxygen will be administered via nasal cannula. Parenteral midazolam and fentanyl will be titrated to patient comfort. Standard skin sterilization, prepping and draping will be applied to the area. The ultrasound probe will be used to identify the iliopubic eminence (IPE). Only skin will be numbed using 2-3 cc of 2% lidocaine and NO bolus of bupivacaine will be injected.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: PENG Block — The pericapsular nerve group (PENG) block is a novel regional anesthesia technique for providing analgesia after hip fractures and hip arthroplasties.
  Arms: Investigational group ("PENG Block" group)
Drug: Lidocaine — 2-3 cc of 2% lidocaine and NO bolus of bupivacaine will be injected.
  Arms: Control group

SUMMARY:
Total hip arthroplasty (THA) is now the second most common joint replacement surgery in the US due in part to an aging population. Opioid sparing analgesic treatments such as lumbar plexus and femoral nerve blocks are effective but they carry a high risk of undesirable lower limb motor or muscle weakness. Fascia iliaca block, on the other hand, does not consistently provide adequate pain relief. Today, early mobilization, rehabilitation and participation in physical therapy is an integral part of enhanced functional recovery program after THA. Because innervation of the hip joint is complex and preservation of lower extremity motor function is paramount, optimal regional analgesic intervention for THA has yet to be defined. The pericapsular nerve group (PENG) block is a novel regional anesthesia technique for providing analgesia after hip fractures and hip arthroplasties. Quality of recovery scores are patient reported outcome measures evaluating recovery after surgery and anesthesia. The quality of recovery-15 (QoR-15) is a validated questionnaire to assess postoperative recovery. The aim of this single center, double blind, randomized controlled trial is to confirm the efficacy of the PENG block for postoperative recovery after primary THA.

Methods: The participants will be randomly assigned to either PENG block group or "no Block" group using a random number generator. The patient will be blinded to the group allocated. The primary outcome will be the quality of recovery 15 score (QoR-15). The secondary outcomes will be visual analog scale score of pain postoperatively, opioid requirements in first 24 hours, ambulation distance on postoperative day1 and patient satisfaction. Statistical analysis will be performed using the student's t-test, Mann-Whitney U test, and Fisher's exact test as appropriate per sample. A p-value of less than 0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
As the practice of anesthesiology has grown increasingly safe, the focus has shifted to improving quality, as evidenced by the robust spread of Enhanced Recovery after Surgery protocols. The implications from poor quality recovery is vast, including prolonged stay in the recovery room or hospital. The Quality of Recovery (QoR-15) questionnaire is a method to measure five dimensions using 15 questions: physical independence, pain, comfort, patient support, emotional state. It is an extensively validated measure of patient-assessed quality of recovery after surgery, having been demonstrated over a variety of clinical settings. QoR-15 scores range from 0 (extremely poor quality of recovery) to 150 (excellent). Mean time to complete the 15-question survey is 3 minutes, a marker of its clinical utility. As we aim to improve our perioperative care and develop approaches to improve medicine in this regard, the QoR-15 provides a useful tool.

The effective postoperative analgesia is vital as acute surgical pain is a potential risk factor for future chronic pain. Persistent pain after THA (more than three months) is reported in 27% of patients and is reported to be correlated with the intensity of early postoperative pain rather than preoperative pain levels. Utilizing regional anesthesia helps to limit the use of opioids, however, which technique is best has yet to be determined. The lumbar plexus blocks, lumbar epidurals, and femoral nerve blocks have been associated with motor weakness. Fascia iliaca compartment block (FICB) has not been found to predictably decrease pain intensity or opioid use. Quadratus lumborum (QL) block is a relatively new regional block found to provide effective analgesia after primary THA, but it can indirectly block lumbar plexus branches and may cause some motor weakness. It is also a deep block and therefore contraindicated in patients on anticoagulation.

Recent anatomic studies confirmed the innervation of the anterior capsule of hip joint to be the obturator nerve, accessory obturator nerve, and femoral nerve. These studies also evaluated the relationship with these nerves and other bony or soft tissue landmarks visible by ultrasound guidance. Previous studies have found histologically that the anterior capsule has predominantly nociceptive fibers, while the posterior capsule is largely made up of mechanoreceptors. The pericapsular nerve group (PENG) block was introduced to target and block these articular branches providing innervation to the hip. Given the case reports showing the efficacy of PENG blocks for hip fracture surgeries, we sought to investigate the analgesic efficacy of PENG blocks for primary and revision THAs. The PENG block targets only the sensory branches and not the posterior mechanoreceptors; there is a potential motor-sparing effect which is desirable for early ambulation, better physical therapy, and earlier discharge. The effective analgesia and early ambulation provided by such regional anesthesia block may have positive impact on patient's mood, sleep, appetite and overall feeling of well-being. A similar postoperative recovery study protocol has been proposed for anterior quadratus lumborum blocks for THA. It remains unclear whether PENG block provides sufficient analgesia and improves the quality of post-operative recovery after primary THA.

The ideal regional anesthesia technique for THA will provide adequate postoperative analgesia, reduced opioid requirements, early ambulation and physical independence. The aim of this single center, double blind RCT is to confirm the efficacy of PENG block for postoperative recovery with respect to parameters mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary total hip arthroplasty
* Patients >=18 years of age
* Patients with an American Society of Anesthesiology (ASA) physical status classification of I, II or III
* Primary THA (first THA operation in the patient's lifetime)

Exclusion Criteria:

* Patients with ASA physical status classification 4 or above
* Patients with allergies/intolerances to local anesthetic
* Patients with pre-existing neurologic or anatomic deficits in the lower extremity on the side of the surgical site
* Patients on chronic opioid use or opioid tolerant (The FDA defines a patient as opioid tolerant if for at least 1 week he or she has been receiving oral morphine 60 mg/day; transdermal fentanyl 25 mcg/hour; oral oxycodone 30 mg/day; oral hydromorphone 8 mg/day; oral oxymorphone 25 mg/day; or an equianalgesic dose of any other opioid)
* Poor understanding of English language.
* Patients with coexisting coagulopathy
* Patients that are pharmacologically anticoagulated will be excluded if placement of peripheral nerve block would be contraindicated according to ASRA (American Society for Regional Anesthesia) guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shana Graves, Study Director — UAB shannagraves@uabmc.edu
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Kukreja P, Uppal V, Kofskey AM, Feinstein J, Northern T, Davis C, Morgan CJ, Kalagara H. Quality of recovery after pericapsular nerve group (PENG) block for primary total hip arthroplasty under spinal anaesthesia: a randomised controlled observer-blinded trial. Br J Anaesth. 2023 Jun;130(6):773-779. doi: 10.1016/j.bja.2023.02.017. Epub 2023 Mar 22. PMID 36964012

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Control group participants will be transferred to the block area preoperatively, and care will proceed as if they were receiving injection.
  Patients will be placed in the supine position resting comfortably. Standard noninvasive monitors will be applied, and oxygen will be administered via nasal cannula. Parenteral midazolam and fentanyl will be titrated to patient comfort. Standard skin sterilization, prepping and draping will be applied to the area. The ultrasound probe will be used to identify the iliopubic eminence (IPE). Only skin will be numbed using 2-3 cc of 2% lidocaine and NO bolus of bupivacaine will be injected.
  Lidocaine: 2-3 cc of 2% lidocaine and NO bolus of bupivacaine will be injected.
Period: Overall Study
Arm/Group | Investigational Group ("PENG Block" Group) | Control Group
Started | 61 | 61
Completed | 56 | 56
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Group ("PENG Block" Group) | Control Group | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 56 | 112
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: YEARS] | 58.5 (14.9) | 62.1 (10.7) | 60.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 64
  Male | 26 | 22 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 28 | 48
  White | 36 | 28 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Recovery After Total Hip Arthroplasty
Description: The quality of recovery-15 is a validated questionnaire to assess postoperative recovery. I Scale is based on 15 questions, each question score range is 0-10 (0 being poor and 10 being excellent) The survey will be conducted at 24 hours after surgery Total score range is 0-150, where a score of 0 would be the worst possible score, and 150 would be the best possible score.
Time Frame: 24 hours after surgery
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Investigational Group ("PENG Block" Group) | Control Group
Number analyzed (Participants) | 56 | 56
score on a scale | 131.5 [116 to 138] | 103 [97 to 111]

2. Secondary Outcome: Evaluating Recovery After Total Hip Arthroplasty
Description: Quality of recovery (QoR) survey at 48 hours after surgery. QoR-15 scores range from 0 (extremely poor quality of recovery) to 150 (excellent quality of recovery).
Time Frame: 2 days after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Investigational Group ("PENG Block" Group) | Control Group
Number analyzed (Participants) | 56 | 56
score on a scale | 136 [22.5 to 143] | 108 [100 to 119.5]

3. Secondary Outcome: Average Pain Medicine Required After Surgery.
Description: Measuring the average milligrams of oral morphine equivalent (OME) consumption at 24 and 48 hours after surgery
Time Frame: 24 and 48 hours after surgery
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Investigational Group ("PENG Block" Group) | Control Group
Number analyzed (Participants) | 56 | 56
Milligrams
  24 hour | 37.3 (29.7) | 59.5 (43.4)
  48hour | 47.1 (40.5) | 75.4 (57.8)

4. Secondary Outcome: Pain Scores After Surgery
Description: Pain scores (visual analog scores VAS) in recovery (PACU), 6, 12, 24 and 48 hours after surgery
Time Frame: Recovery (PACU), 6, 12, 24 and 48 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Group ("PENG Block" Group) | Control Group
Number analyzed (Participants) | 56 | 56
score on a scale
  PACU | 1.8 (1.5) | 2.3 (1.7)
  6 Hour | 2.3 (2.7) | 2.5 (2.8)
  12 Hour | 1.9 (2.3) | 2.0 (2.3)
  24 Hour | 2.8 (2.3) | 2.8 (2.2)
  48 Hour | 2.0 (1.6) | 2.7 (2.3)

5. Secondary Outcome: Ambulation Distance After Surgery
Description: ambulation distance as recorded by physical therapist at 24 and 48 hours after surgery
Time Frame: 24 and 48 hours after surgery
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Investigational Group ("PENG Block" Group) | Control Group
Number analyzed (Participants) | 56 | 56
feet
  24 Hour | 121.3 (75.3) | 104.0 (72.0)
  48 Hour | 78.9 (47.5) | 81.2 (52.0)

6. Secondary Outcome: Total Patients Using Antiemetics After Surgery
Description: use of any medication for nausea or vomiting prevention after surgery
Time Frame: up to 2 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Group ("PENG Block" Group) | Control Group
Number analyzed (Participants) | 56 | 56
Participants | 17 | 19

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Investigational Group ("PENG Block" Group) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT04591353/Prot_SAP_001.pdf